CLINICAL TRIAL: NCT05337748
Title: Clinical Validation of the Lexie Lumen Over the Counter Hearing Aid
Brief Title: Clinical Validation of the Lexie Lumen Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hearX Group (Industry)
Collaborators: University of Pretoria (Other)
Responsible Party: Principal Investigator, De Wet Swanepoel, Principal Investigator, hearX Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LexieLumen
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aid; hearing rehabilitation; self-fitting hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: The experimental group will undergo the self-test and fitting (Lexie STF) intervention and the experimental group will undergo the professional test and fit (Lexie PTF) intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental : Lexie Self Test and Fit Group (Lexie STF) (Experimental): The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with a slimtube and dome. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing check (pure tones presented via the hearing aids). The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
  Interventions: Device: Lexie Self Test and Fit Group
- Control: Lexie Professional Test and Fit Group (Lexie PTF) (Active Comparator): The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with slimtube and dome. Hearing aids will be fitted by a certified audiologist according to a gold-standard prescriptive formula (NAL-NL2) using a clinically obtained diagnostic pure tone audiogram. Participants will have access to the smartphone application, but the settings will be limited with only options to change the volume of the hearing aids.
  Interventions: Device: Lexie Professional Test and Fit Group

INTERVENTIONS:
Device: Lexie Self Test and Fit Group — The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with a slimtube and dome. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing check (pure tones presented via the hearing aids). The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
  Other Names: Lexie STF)
  Arms: Experimental : Lexie Self Test and Fit Group (Lexie STF)
Device: Lexie Professional Test and Fit Group — The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with slimtube and dome. Hearing aids will be fitted by a certified audiologist according to a gold-standard prescriptive formula (NAL-NL2) using a clinically obtained diagnostic pure tone audiogram. Participants will have access to the smartphone application, but the settings will be limited with only options to change the volume of the hearing aids.
  Other Names: Lexie PFT
  Arms: Control: Lexie Professional Test and Fit Group (Lexie PTF)

SUMMARY:
More than half a billion people globally have hearing loss. Most hearing loss is sensorineural, meaning that the hearing loss is irreversible and requires rehabilitation. The majority of people with hearing loss have mild to moderate degrees, for which the most effective treatment options are hearing aids. Over the past few years, there have been many developments in hearing technology and the service delivery models in which they are supplied. Traditional hearing care models include several visits to a qualified hearing professional who must both perform diagnostics and prescribe hearing aids, which in the past has been the only way to obtain hearing aids. However, newer developments include forms of self-fitting hearing aids that enable a user to perform threshold measurements to determine the degree of hearing loss and automatically program and fine-tune hearing aids. These devices are now becoming available as direct-to-consumer (DTC) or over-the-counter (OTC) hearing aids. Furthermore, alternative care models have been suggested to bolster access and uptake of assistive technology for hearing loss. Regulations on DTC and OTC hearing aids are starting to come into effect. In 2017, the FDA Reauthorization Act of 2016 directed the FDA to create a category for OTC hearing aids for adults with perceived mild-to-moderate hearing loss. In October 2021, the FDA formally proposed a rule to establish the OTC hearing aid category as part of this process. These changes in regulations would mean that soon, many of these self-fitting devices will become available. In response to these changes in service delivery models, the hearX group recently developed the Lexie Lumen hearing aids that can perform in-situ hearing threshold estimations and automatically prescribe hearing aid gain settings that closely approximate the gold-standard NAL-NL2 fitting prescription. This study aims to evaluate whether the performance of the novel Lexie self-test and self-fitting hearing aid is equivalent to the same hearing aid programmed professionally by an audiologist using a professionally obtained audiogram.

DETAILED DESCRIPTION:
Objective: To examine the difference in outcomes (satisfaction and objective benefit) of the Lexie self-test and self-fitting (Lexie- STF) hearing aid versus a Lexie hearing aid fitted professionally with a clinically obtained audiogram (Lexie-PTF) (n = 60).

Hypothesis: It is hypothesized that the Lexie-STF (experimental group) will be non-inferior to the Lexie-PFT (control group) in terms of perceived satisfaction, speech perception in noise and real-ear measurements.

Design: A randomized control trial (RCT) will be conducted cross-sectionally (45 days) to evaluate the efficacy of Lexie-STF compared to Lexie-PTF.

Setting: This study will involve clinical, audiometric testing as well as a user field-trial of the fitted hearing aids.

Participants: Eligible participants will include 60 adults (18 to 99 years) with a self-perceived level of hearing loss, free from symptoms of ear disease or excessive cerumen and who own a smartphone (Android or iOS). Participants will be recruited for each group and will randomly be assigned using a computer-generated randomization by an independent research assistant, after being stratified for sex and degree of hearing loss.

Intervention: The experimental group (Lexie-STF) will be provided with Lexie Lumen hearing aids and accompanying smartphone application, that will be automatically fitted according to the participants in-situ audiogram. Participants will then be able to self-adjust their hearing aid settings (prescriptive gain) after a period of two weeks. The control group (Lexie PTF) will be professionally fitted by a certified audiologist with the Lexie Lumen hearing aids, according to gold-standard NAL-NL2 prescriptive gain targets using a standard clinically obtained audiogram.

Outcome measures: The main outcome measure is the Abbreviated Profile of Hearing Aid Benefit (APHAB). Secondary outcome measures will be the International Outcome Inventory for Hearing Aids (IOI-HA), the QuickSIN speech-in-noise test and real-ear-measurements (REMs).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between the ages of 18 to 99 years, living in South Africa.
2. Good English proficiency (measured using an online English proficiency test as well as self-report of English speaking competence)
3. Must have a self-perceived hearing loss
4. Mild to severe sensorineural hearing loss (thresholds <= 80 dB HL across frequencies bilaterally)
5. Possession of a smartphone compatible with the Lexie app (iOS or Android)
6. Access to mobile data to operate the Lexie app.
7. Willingness and availability to participate in the study over a period of 45 days

Exclusion Criteria:

1. Normal hearing or profound hearing loss
2. Active outer or middle ear disease
3. Poor English proficiency
4. Diagnosed cognitive impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: De Wet Swanepoel, PhD, Principal Investigator — hearX Group
Locations (1):
- University of Pretoria, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chadha S, Kamenov K, Cieza A. The world report on hearing, 2021. Bull World Health Organ. 2021 Apr 1;99(4):242-242A. doi: 10.2471/BLT.21.285643. No abstract available. PMID 33953438
- [Background] Keidser G, Convery E. Self-Fitting Hearing Aids: Status Quo and Future Predictions. Trends Hear. 2016 Apr 12;20:2331216516643284. doi: 10.1177/2331216516643284. PMID 27072929
- [Derived] De Sousa KC, Manchaiah V, Moore DR, Graham MA, Swanepoel W. Effectiveness of an Over-the-Counter Self-fitting Hearing Aid Compared With an Audiologist-Fitted Hearing Aid: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Jun 1;149(6):522-530. doi: 10.1001/jamaoto.2023.0376. PMID 37052929

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental : Lexie Self Test and Fit Group (Lexie STF): The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with a slimtube and dome. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing check (pure tones presented via the hearing aids). The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
  Lexie Self Test and Fit Group: The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing test. The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms.
Period: Overall Study
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Started | 35 | 33
Completed | 33 | 33
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Originally, 68 participants met the inclusion criteria for the study. In the Lexie STF group, 1 participant was lost to follow up and one discontinued the intervention. For analysis, one participant was excluded from this group due to an incorrect fitting resulting from researcher error. In the Lexie PTF group, 33 participants met the inclusion criteria, but one was excluded from analysis at the end of the study to not being matched to target and experiencing significant device feedback.
Groups:
- Experimental : Lexie Self Test and Fit Group (Lexie STF): The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing test. The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
  Lexie Self Test and Fit Group: The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with a slimtube and dome. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing check (pure tones presented via the hearing aids). The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
- Total: Total of all reporting groups
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF) | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (13.1) | 65.3 (14.9) | 63.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 15 | 18 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27 | 22 | 49
  Race: Black | 2 | 1 | 3
  Race: Asian | 2 | 9 | 11
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 32 | 32 | 64
Pure tone audiometry [Mean (Standard Deviation); unit: Decibel Hearing Level (dB HL)] | 38.4 (11.7) | 41.8 (13.6) | 40.1 (25.3)

OUTCOME MEASURES:

1. Primary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The Abbreviated Profile of Hearing Aid Benefit (APHAB) is a 24 item self-assessment inventory in which patients report the amount of trouble they experience hearing and communicating in noise in different everyday listening environments. Benefit is calculated by comparing the patient's reported difficulty in the unaided condition with their amount of difficulty when using amplification. The APHAB produces scores for 4 subscales: Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV).The final score is determined by subtracting the aided average from the unaided average, keeping in mind that the score indicates how frequently the individual experiences communication difficulty. Therefore a higher score indicates a poorer outcome. (Minimum score 1% to a maximum score of 99%).
Time Frame: Change from baseline assessment to final assessment after 30 day field trial use.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale (1-99)
Groups:
- Experimental : Lexie Self Test and Fit Group (Lexie STF): The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids. Participants will self-perform an in-situ hearing test and prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds. Participants will be fitted according to the customized, Lexie optimal fit prescribed gain setting. The optimal settings include the original gain and compression requirements that NAL-NL2 suggests for various audiograms. No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
  Lexie Self Test and Fit Group: The intervention offered is a hearing aid fitting with Lexie Lumen hearing aids coupled with a slimtube and dome. The hearing aids will be accompanied and operated using the Lexie smartphone application. Participants will self-perform an in-situ hearing check (pure tones presented via the hearing aids). The prescriptive gain of the hearing aids will be programmed and applied automatically using the obtained in-situ hearing thresholds No additional band equalizer or compression adjustments are added. After a specified period of time, participants will be able to self-adjust the hearing aids using the smartphone application.
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Number analyzed (Participants) | 32 | 32
score on a scale (1-99) | 30.1 (21.9) | 21.4 (21.5)

2. Secondary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA)
Description: IOI HA is a seven item questionnaire designed to evaluate effectiveness of hearing aid treatment. The responses of the items are assigned a value of 1 to 5, with higher scores indicating a more favorable outcome. The total score is calculated as the sum of all the subscales. Minimum score for the total score is 7 and maximum score 35.
Time Frame: Final assessment after 30 day field use
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale (7-35)
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Number analyzed (Participants) | 32 | 32
score on a scale (7-35) | 31 [30 to 33] | 31 [28 to 34]

3. Secondary Outcome: QuickSIN Speech in Noise Test
Description: The QuickSIN measures a persons ability to accurately hear speech in noise by determining a signal-to-noise ratio loss. A list of six sentences with five key words per sentence is presented in four-talker babble noise. The sentences are presented at pre-recorded signal-to-noise ratios which decrease in 5-dB steps from 25 (very easy) to 0 (extremely difficult). To score, the number of correctly repeated words from each of the six sentences are counted. The SNR loss is calculated by subtracting the total number of correct words from 25.5. Three lists are averaged to obtain an average SNR score. The SNRs used are: 25, 20, 15, 10, 5 and 0, encompassing normal to severely impaired performance in noise. Benefit scores are calculated as unaided (without hearing aids) -aided (with hearing aids) score. Benefit scores at 30 days are presented in the data table.
Time Frame: Baseline and benefit at the end of 30 day field use
Population: Originally,68 participants met the inclusion criteria for the study. In the Lexie STF group, 1 participant was lost to follow up and one discontinued the intervention. For analysis, one participant was excluded from this group due to an incorrect fitting resulting from researcher error. In the Lexie PTF group, 33 participants met the inclusion criteria, but one was excluded from analysis at the end of the study to not being matched to target and experiencing significant device feedback.
Measure: Mean (Standard Deviation); unit: Decibel Signal to Noise Ratio (dB SNR)
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Number analyzed (Participants) | 32 | 32
Decibel Signal to Noise Ratio (dB SNR) | 1.6 (4.4) | 3.5 (4.5)

4. Secondary Outcome: Digits-in-noise Test (DIN)
Description: The DIN measure primarily the auditory, or bottom-up, speech recognition abilities in noise. The test determines a speech reception threshold by presenting spoken digit triplets (e.g., 3-4-7) in speech weighted background masking noise. Twenty three digits are presented adaptively at different signal to noise ratios, based on correct or incorrect recognition of the digits. The speech reception threshold is determined by averaging the signal to noise ratios of the last 19 digit triplets. Benefit scores are calculated as unaided baseline- aided at 30 days after field trial use. Benefit scores are presented in the data table.
Time Frame: Baseline unaided test and aided fitting final assessment after 30 day field use
Population: 68 participants met the inclusion criteria for the study. In the Lexie STF group, 1 participant was lost to follow up and one discontinued the intervention. For analysis, one participant was excluded from this group due to an incorrect fitting resulting from researcher error. In the Lexie PTF group, 33 participants met the inclusion criteria, but one was excluded from analysis at the end of the study to not being matched to target and experiencing significant device feedback.
Measure: Mean (Standard Deviation); unit: Decibel Signal to Noise Ratio (dB SNR)
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Number analyzed (Participants) | 32 | 32
Decibel Signal to Noise Ratio (dB SNR) | .50 (2.6) | 0.13 (4.7)

5. Secondary Outcome: Live Speech Mapping Using Real Ear Measurements (REM)
Description: Real Ear Measurements (REM) involves placing a fine probe microphone into the ear canal to measure the sound at the eardrum. The hearing aid will be inserted in the ear alongside the probe microphone to measure the amplification effect within the patients ear taking into account the patient ear acoustics. Adjustments to the hearing aid can be made and measurement to best match the prescription target. The specific REM measure used will be Live Speech Mapping, which assesses the hearing aid output using realistic speech presented via a loudspeaker with the hearing aid in its normal mode of operation. The outcome measure of Live Speech Mapping is the decibel sound pressure level (dB SPL) across a range of frequencies (250Hz to 4000Hz), calculated as the difference from the NAL-NL2 target (i.e. NAL-NL2 target- measured dB SPL).
Time Frame: Final assessment after 30 day field use
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: dB SPL
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
Number analyzed (Participants) | 32 | 32
dB SPL
  250Hz | 0.6 (2.5) | 3.0 (4.1)
  500Hz | 1.3 (3.1) | 2.7 (4.0)
  1000 Hz | 4.7 (6.2) | 4.3 (6.4)
  2000 Hz | -2.7 (6.8) | 0.6 (6.5)
  4000 Hz | 6.9 (7.6) | 4.4 (6.4)

ADVERSE EVENTS:
Time Frame: 5.5 months
Description: Any unexpected medical occurrence, unintended disease, injury, or clinical signs in subjects, users or other persons related to the investigational medical device.
Arm/Group | Experimental : Lexie Self Test and Fit Group (Lexie STF) | Control: Lexie Professional Test and Fit Group (Lexie PTF)
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT05337748/Prot_SAP_001.pdf